CLINICAL TRIAL: NCT03160872
Title: Ovarian Reserve Does Not Predict Pregnancy in Non-Infertile Women: An Assessment Using the Donor Sperm Insemination Model
Brief Title: Anti-Müllerian Hormone is Not Predictive of Pregnancy in Donor Insemination Cycles in Non-infertile Women
Status: Completed | Type: Observational
Sponsor: Fundacion Dexeus (Other)
Responsible Party: Principal Investigator, Iñaki González Foruria, MD., Fundacion Dexeus
Other Study IDs: SMD-2016-033
Record Dates: First submitted 2017-05-18; First posted 2017-05-19 (Actual); Last update posted 2017-05-19 (Actual); Status verified 2017-05

CONDITIONS: Infertility
Keywords: Donor sperm insemination; Anti Mullerian Hormone; Ovarian reserve; Antral follicle count
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Women who undergo donor sperm insemination: Non infertile women who undergo donor sperm insemination cycle
  Interventions: Diagnostic Test: Anti Mullerian Hormone Measurement

INTERVENTIONS:
Diagnostic Test: Anti Mullerian Hormone Measurement — Anti Mullerian Hormone was measured in all patients within two months before the first insemination cycle

SUMMARY:
To evaluate if ovarian reserve (measured by means of anti-mullerian hormone -AMH- and antral follicle count -AFC-) can predict pregnancy in donor insemination cycles (dIUI) performed in non-infertile women.

ELIGIBILITY:
Inclusion Criteria:

* absence of male partner
* complete azoospermia or the presence of a genetic condition in the partner that made the couple opt for donor sperm
* absence of previous history of infertility.
* d ta on AMH and AFC assessment before the first dIUI cycle.

Exclusion Criteria:

* previous history of infertility.
* Presence of any gynaecological condition that could impair the inseminations results:

  * endometriosis, hydrosalpinx,…

Ages: 18 Years to 43 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Non Infertile women who undergo a donor sperm insemination due to absence of male partner or complete azoospermia or the presence of a genetic condition in the partner that made the couple opt for donor sperm.
Sampling Method: Probability Sample
Enrollment: 143 (Actual)
Dates: Start 2013-01-01 (Actual); Primary Completion 2016-06-30 (Actual); Study Completion 2016-12-15 (Actual)

PRIMARY OUTCOMES:
Clinical Pregnancy | 6 weeks after insemination procedure
  Clinical Pregnancy evaluated by ultrasound with fetal heart beat

SECONDARY OUTCOMES:
Miscarriage rate | Evaluated until 15 weeks after insemination procedure
  Number of clinical miscarriage after clinical pregnancy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Catteau-Jonard S, Roux M, Dumont A, Delesalle AS, Robin G, Dewailly D. Anti-Mullerian hormone concentrations and parity in fertile women: the model of oocyte donors. Reprod Biomed Online. 2017 May;34(5):541-545. doi: 10.1016/j.rbmo.2017.02.010. Epub 2017 Mar 1. PMID 28285954
- [Background] Hvidman HW, Bentzen JG, Thuesen LL, Lauritsen MP, Forman JL, Loft A, Pinborg A, Nyboe Andersen A. Infertile women below the age of 40 have similar anti-Mullerian hormone levels and antral follicle count compared with women of the same age with no history of infertility. Hum Reprod. 2016 May;31(5):1034-45. doi: 10.1093/humrep/dew032. Epub 2016 Mar 9. PMID 26965431
- [Background] Somigliana E, Lattuada D, Colciaghi B, Filippi F, La Vecchia I, Tirelli A, Baffero GM, Paffoni A, Persico N, Bolis G, Fedele L. Serum anti-Mullerian hormone in subfertile women. Acta Obstet Gynecol Scand. 2015 Dec;94(12):1307-12. doi: 10.1111/aogs.12761. Epub 2015 Sep 16. PMID 26332870
- See also: Related Info — http://www.dexeus.com